CLINICAL TRIAL: NCT03045744
Title: Long-term Paired Associative Stimulation in Rehabilitation of Spinal Cord Injury Patients
Brief Title: Long-term PAS in Rehabilitation After SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Validia Rehabilitation (Unknown); University of Helsinki (Other)
Responsible Party: Principal Investigator, Anastasia Shulga, Principle Investigator, Helsinki University Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ULD 8100014
Record Dates: First submitted 2017-02-02; First posted 2017-02-07 (Estimated); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- incomplete SCI patients (Experimental)
  Interventions: Device: long-term paired associative stimulation

INTERVENTIONS:
Device: long-term paired associative stimulation — Paired associative stimulation (PAS) administered 3 times per week. PAS comprises transcranial magnetic stimulation (eXimia magnetic stimulator, Nexstim Ltd, Helsinki, Finland) and peripheral nerve stimulation (given with Dantec Keypoint® electroneuromyography device (Natus Medical Incorporated, Pleasanton, CA, USA)).

SUMMARY:
The investigators have recently shown in two pilot incomplete SCI patients that long-term paired associative stimulation is capable of restoring voluntary control over some paralyzed muscles and enhancing motor output in the weak muscles (1). In this study, the investigators will administer long-term paired associative stimulation to incomplete SCI patients in a long-term manner, keeping each patient in the study for as long as continuous improvement is observed.

ELIGIBILITY:
Inclusion Criteria:

* incomplete SCI

Exclusion Criteria:

* epilepsy
* metal inclusion in the head area
* pacemaker
* hearing device
* high intracranial pressure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Daniels and Worthingham's Muscle Testing | 2 days after the last stimulation session
Daniels and Worthingham's Muscle Testing | 1 month after the last stimulation session

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia Shulga, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- BioMag laboratory, Helsinki University Central Hospital, Helsinki, Uusimaa, Finland

REFERENCES:
- [Result] Rodionov A, Savolainen S, Kirveskari E, Makela JP, Shulga A. Restoration of hand function with long-term paired associative stimulation after chronic incomplete tetraplegia: a case study. Spinal Cord Ser Cases. 2019 Oct 1;5:81. doi: 10.1038/s41394-019-0225-5. eCollection 2019. PMID 31632739
- [Result] Holopainen K, Tolmacheva A, Bersch I, Haakana P, Pohjonen M, Kirveskari E, Arokoski J, Shulga A. Stable improvement in hand muscle strength in incomplete spinal cord injury patients by long-term paired associative stimulation-a case series study. Front Neurol. 2025 Feb 4;16:1486591. doi: 10.3389/fneur.2025.1486591. eCollection 2025. PMID 39968455